CLINICAL TRIAL: NCT07059806
Title: T1CARE: A Randomized Trial of a Novel Intervention to Address Social Determinants of Health in Young Adults With Type 1 Diabetes
Brief Title: T1CARE: A Trial of a Novel Intervention to Address Social Determinants of Health in Young Adults With Type 1 Diabetes
Acronym: T1CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000040438; 1R01DK139558-01A1 (NIH)
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Participants will complete a standardized Social Determinants of Health (SDOH) screening.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T1CARE (Experimental): Patients who are randomized to the intervention arm will be contacted by the Community Health Navigator (CHN) from Project Access-New Haven (PA-NH) (PA-NH). The CHN will conduct an in-depth in-person intake interview to understand the patient's social and clinical need. Additional assessment will include access to insulin, diabetes technologies, and other supplies. The intake will be the basis for a personalized intervention that will respond to patient's unique needs. The initial interview will be audio-recorded to allow for qualitative data analysis. Outcomes will be measured at 6 months. Participants in the T1CARE group will have an option to join a social media platform in addition to receiving individualized support from the CHN.
  Interventions: Behavioral: T1CARE
- Standard Care (No Intervention): Participants in the control group will be receive standard screening for SDOH and standard diabetes care at their respective clinics.

INTERVENTIONS:
Behavioral: T1CARE — The intervention includes navigation by a Community Health Navigator (CHN), who will assess and help address patients' SDOH-related needs, coordinate care, and provide social support.
  Arms: T1CARE

SUMMARY:
Randomized controlled trial with a wait list control arm. Participants will be randomized 1:1 to T1CARE or wait list usual care arm. Participants will be recruited from the Yale Adult and Pediatric Diabetes Centers. Patients assigned to T1CARE will receive support from a Community Health Navigator at Project Access-New Haven.

DETAILED DESCRIPTION:
Primary Objective To determine whether the T1CARE intervention improves resolution of health-related social needs compared to usual care.

Secondary Objectives

1. To assess the feasibility and acceptability of the T1CARE intervention.
2. To evaluate the impact of T1CARE on patient-reported outcomes, including diabetes distress, illness intrusiveness, and quality of life.
3. To examine preliminary effects on clinical outcomes, particularly changes in HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes
* fluent in Spanish or English who reside in the greater New Haven area

Exclusion Criteria:

* cognitive impairment and otherwise unable to give written informed consent about participating in this study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with resolution of health-related social needs | 6 months
  Resolution of health-related social needs, assessed via adapted Accountable Health Communities (AHC) Model screening questions. Yes/No for resolution.

SECONDARY OUTCOMES:
Mean score Diabetes Distress Scale (T1-DDS) | 6 months
  The T1-DDS is a 28-item self-report instrument. Each item is rated on a 6-point scale from (1) "not a problem" to (6) "a very significant problem." Total score range 1-6 with higher scores indicating more distress. Investigators will analyze between-group change of the within-group change.
Mean score Illness intrusiveness rating scale (IIRS) | 6 months
  IIRS comprised of 13 items that ask patients to rate the degree to which their "illness and/or its treatment" interfere with life domains central to quality of life. Total score range 13 to 91, with higher scores indicating greater illness intrusiveness. Investigators will analyze between-group change of the within-group change.
Mean score DAWN Impact of Diabetes Profile (DIDP) scale | 6 months
  Quality of life measured by the brief (7 item) DIDP scale (DAWN Impact of Diabetes Profile). Total score range 1-7 with higher scores indicating more negative impact. Investigators will analyze between-group change of the within-group change.
Mean score Patient satisfaction survey | 6 Months
  Patient satisfaction with the intervention will be assessed with 2 questions on a 5-point Likert scale that address whether they were satisfied and would recommend the approach used for their care (which could have been T1CARE or usual care alone) to other patients. Total score range 1-5, higher scores indicate more satisfaction.
Change in HbA1c | 6 months
  Change in HbA1c at baseline and 6 months. Investigators will analyze between-group change of the within-group change.

CONTACTS AND LOCATIONS:
Overall Officials: Kasia Lipska, MD, MHS, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale Adult Diabetes Center, New Haven, Connecticut
  - Yale Children's Diabetes Center, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
Metadata associated with the datasets will be submitted to the NIDDK repository or Vivli.
Time Frame: Scientific data will be shared as soon as possible. Scientific data included in published manuscripts will be available at time of publication. All other data generated will be shared no later than the end of the award. Study data will be stored for 10 years (this is Vivli's policy).
Access Criteria: * Health/Medical/Biomedical - The dataset can only be used for studying health, medical, or biomedical conditions and does not include the study of population origins or ancestry.
  * IRB Approval Required (IRB) - The requesting institution's IRB or equivalent body must approve the requested use.